CLINICAL TRIAL: NCT00721630
Title: Phase II Study of a Novel Capecitabine Dosing Schedule in Combination With Lapatinib, Based on the Norton-Simon Mathematical Method in Patients With HER2 Overexpressed/Amplified, Trastuzumab (Herceptin) -Refractory, Metastatic Breast Cancer
Brief Title: Novel Capecitabine Dosing Schedule in Combination With Lapatinib, Based on the Norton-Simon Mathematical Method in Patients With HER2 Overexpressed/Amplified, Trastuzumab (Herceptin) -Refractory, Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-025
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Results first posted 2017-08-15 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2016-07

CONDITIONS: Breast Cancer
Keywords: CAPECITABINE; LAPATINIB
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Lapatinib

ARMS (1):
- 1 (Experimental): The regimen consists of capecitabine 2,000mg twice daily for 7 days followed by a 7-day rest in combination with lapatinib 1,250mg orally daily.
  Interventions: Drug: capecitabine, lapatinib

INTERVENTIONS:
Drug: capecitabine, lapatinib — Capecitabine 2,000mg twice daily for 7 days followed by a 7-day rest in combination with lapatinib 1,250mg orally daily. Cycle length is 28 days (+/- 2 days).Toxicity assessment will occur q2 weeks for the first 4 weeks, then q4 weeks(+/- 2 days). Radiographic response assessment will take place q12 weeks (+/- 1 week). LVEF assessment will be repeated q12 weeks (+/- 1 week).

SUMMARY:
HER2 is a protein that sits on the surface of breast cancer cells in some people. Because you are one of these people, your breast cancer is called "HER2-positive." The HER2 protein is involved in the growth of your breast cancer. Certain drugs can interfere with the ability of the HER2 protein to cause breast cancer growth. Trastuzumab is one of these drugs. You must have already received trastuzumab as treatment for your breast cancer to be considered for this study.

Other drugs are being studied in women with HER2-positive breast cancer. Lapatinib (Tykerb™) blocks signals that stimulate HER2-positive breast cancers to grow. The FDA approved lapatinib for use with capecitabine (Xeloda™) in patients who have metastatic breast cancer that has grown or spread after treatment with trastuzumab.

Capecitabine was approved by the FDA in 1998 for treating metastatic breast cancer. Capecitabine is a pill that blocks the way cancer cells multiply and grow. Usually, this medicine is taken twice a day for fourteen days. Then, patients do not take the pill for seven days. With this schedule and dose, some patients have had side effects that interfered with their comfort. We have used mathematical models to recommend a new schedule of capecitabine. In animals, 7 days of treatment with capecitabine followed by a 7-day break was safer and more active against breast cancer. The purpose of this study is to find out what effect (both good and bad) capecitabine has on you and your breast cancer when given in this new schedule and combined with lapatinib.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of invasive adenocarcinoma of the breast confirmed by histology or cytology at MSKCC.
* Clinical evidence of metastatic breast cancer.
* HER2 overexpression and/or amplification as determined by immunohistochemistry (3+) or FISH (≥2.0).
* Progressive disease following treatment with trastuzumab for metastatic breast cancer or as adjuvant therapy (either single-agent or combination therapy)
* Prior therapy inclusion:

  * No more than two prior chemotherapy regimens allowed for advanced stage disease
  * No prior fluoropyrimidine in the metastatic setting. Adjuvant fluoropyrimidine is permitted if >6 months prior to treatment on study.
  * No restriction for prior hormonal therapy. No concurrent use of endocrine therapy is permitted.
  * No more than 450mg/m2 cumulative dose of prior doxorubicin
  * At least 3 weeks since prior chemotherapy or radiation therapy
* Age ≥ or = to 18. Because no dosing or adverse event data are currently available on the use of lapatinib in patients <18 years of age, children are excluded from this study.
* Patients must be willing to discontinue sex hormonal therapy e.g., birth control pills, ovarian hormonal replacement therapy, etc., prior to enrollment. Women of childbearing potential must be willing to consent to using effective contraception while on treatment and for a reasonable period thereafter.
* Negative HCG pregnancy test for premenopausal women of reproductive capacity and for women less than 12 months after the menopause.
* Asymptomatic, central nervous system metastases are permitted if patients remain clinically stable after discontinuation of corticosteroids and anticonvulsants.
* ECOG performance status < or = to 2
* Life expectancy of greater than 12 weeks

Patients must have normal organ and marrow function as defined below:

* leukocytes ≥ or = to 3,000/μL
* absolute neutrophil count ≥ or = 1,500/μL
* platelets ≥ or = 100,000/μL
* total bilirubin within normal institutional limits AST (SGOT)/ALT(SGPT) ≤ or = 2.5x institutional upper limit of normal serum creatinine within normal institutional limits

  * Cardiac ejection fraction at or above the lower limit of normal of 50% as measured by multigated radionuclide angiography (MUGA) scan. If LVEF is greater than 70%, and ECHO should be performed as well. Baseline and on treatment scans should be performed using the same modality and preferably at the same institution.
  * Ability to understand and the willingness to sign a written informed. consent document.
  * Able to swallow and retain oral medication.

Exclusion Criteria:

* Patients may not be receiving any concurrent anticancer therapy or investigational agents with the intention of treating breast cancer.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to lapatinib or capecitabine.
* Known DPD deficiency.
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within 6 months of study entry, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because lapatinib is member of the 4- anilinoquinazoline class of kinase inhibitors with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with lapatinib, breastfeeding should be discontinued if the mother is treated with lapatinib.
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with lapatinib. Appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated.
* Patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption,uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis).
* Concomitant requirement for medication classified as CYP3A4 inducers or inhibitors:
* Medications that inhibit or induce CYP3A4 are prohibited. Eligibility of patients receiving medications or substances known to affect, or with the potential to affect the activity or pharmacokinetics of lapatinib will be determined following review of their use by the Principal Investigator.
* Renal function as measured by creatinine clearance < 30ml/min
* Patients are permitted to participate in other non-therapeutic clinical trials while receiving treatment on this study (ie, experimental imaging, minor procedures necessary for tissue acquisition on study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Traina, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan-Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York
  - Memorial Sloan-Kettering Cancer Center at Phelps Memorial Hospital Center, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual 7/10/2008, Protocol Closed to Accrual 7/27/2010, Primary Completion Date 7/14/2016, Recruitment location is the medical clinic
Groups:
- Capecitabine + Lapatinib: The regimen consists of capecitabine 2,000mg twice daily for 7 days followed by a 7-day rest in combination with lapatinib 1,250mg orally daily.
  capecitabine, lapatinib: Capecitabine 2,000mg twice daily for 7 days followed by a 7-day rest in combination with lapatinib 1,250mg orally daily. Cycle length is 28 days (+/- 2 days).Toxicity assessment will occur q2 weeks for the first 4 weeks, then q4 weeks(+/- 2 days). Radiographic response assessment will take place q12 weeks (+/- 1 week). LVEF assessment will be repeated q12 weeks (+/- 1 week).
Period: Overall Study
Arm/Group | Capecitabine + Lapatinib
Started | 24
Completed | 23
Not Completed | 1
Not completed — Participant found to be ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Capecitabine + Lapatinib
Number analyzed (Participants) | 24
Age, Continuous [Median (Full Range); unit: years] | 54 [34 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Estimate Efficacy of Capecitabine 7/7 in Combination With Lapatinib in Patients With HER2 Overexpressed/Amplified, Trastuzumab-refractory, Metastatic Breast Cancer as Determined by Overall Response Rate (Complete Response (CR) + Partial Response (PR))
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Capecitabine + Lapatinib
Number analyzed (Participants) | 23
Participants
  Partial Response | 5
  Stable Disease >/= 6 months | 6
  Stable disease <6 months | 11
  Progression of disease | 1

2. Secondary Outcome: Number of Participants With Toxicities Associated With Capecitabine and Lapatinib
Description: Toxicities evaluated according to NCI CTC v.3
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Capecitabine + Lapatinib
Number analyzed (Participants) | 23
Participants | 23

ADVERSE EVENTS:
Arm/Group | Capecitabine + Lapatinib
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 9/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine + Lapatinib (N=23)
ALT (Investigations) | 1
AST (Investigations) | 1
Ataxia (Nervous system disorders) | 2
Confusion (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Glucose, high (Metabolism and nutrition disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
INR (Investigations) | 1
Nausea (Gastrointestinal disorders) | 1
Neurology - Other (Nervous system disorders) | 1
PTT (Investigations) | 1
Limb Pain (Musculoskeletal and connective tissue disorders) | 1
Rash - hand-foot skin (Skin and subcutaneous tissue disorders) | 1
Seizure (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine + Lapatinib (N=23)
Anemia (Blood and lymphatic system disorders) | 5
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 16
Diarrhea (Gastrointestinal disorders) | 19
AST (Hepatobiliary disorders) | 16
Fatigue (General disorders) | 15
ALT (Hepatobiliary disorders) | 12
Nausea (Gastrointestinal disorders) | 12
Alkaline Phosphatase (Investigations) | 11
Vomiting (Gastrointestinal disorders) | 8
Hypoalbuminemia (Metabolism and nutrition disorders) | 7
Dry Skin (Skin and subcutaneous tissue disorders) | 7
Hyperglycemia (Metabolism and nutrition disorders) | 7
Sensory Neuropathy (Nervous system disorders) | 7
Rash/desquamation (Skin and subcutaneous tissue disorders) | 7
White blood cell decreased (Investigations) | 6
Mucositis - oral cavity (Gastrointestinal disorders) | 6
Hypernatremia (Metabolism and nutrition disorders) | 6
Hyperbilirubinemia (Investigations) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Constipation (Gastrointestinal disorders) | 4
Dyspena (Respiratory, thoracic and mediastinal disorders) | 4
Nail changes (Skin and subcutaneous tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Creatinine (Investigations) | 3
Dizziness (Nervous system disorders) | 3
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3
INR (Investigations) | 3
Pain - Back (Musculoskeletal and connective tissue disorders) | 3
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 3
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 2
Cheilitis (Gastrointestinal disorders) | 2
Dermatology/Skin, other (Skin and subcutaneous tissue disorders) | 2
Fever (in the absence of neutropenia) (General disorders) | 2
PTT (Investigations) | 2
Pain - joint (Musculoskeletal and connective tissue disorders) | 2
Pain - Other (General disorders) | 2
Platelets (Investigations) | 2
Potassium, high (Metabolism and nutrition disorders) | 2
Potassium, low (Metabolism and nutrition disorders) | 2
Pruritis/itching (Skin and subcutaneous tissue disorders) | 2
Vaginal dryness (Reproductive system and breast disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes